CLINICAL TRIAL: NCT02406248
Title: A Multicenter, Single Arm, Open Label, Phase IV Study to Evaluate Safety and to Describe the Cumulative Incidence of Major Cardiovascular Events of Ticagrelor in Taiwanese Patients With Non ST-segment Elevation Myocardial Infarction
Brief Title: Brilinta Taiwan Post Approval Safety Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5130C00103
Record Dates: First submitted 2015-03-19; First posted 2015-04-02 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Non ST-elevation Myocardial Infarction
Keywords: NSTEMI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): Ticagrelor 180mg loading dose taken orally, followed by 90mg twice daily (bd)
  Interventions: Drug: Ticagrelor 180mg loading dose taken orally, followed by 90mg twice daily (bd)

INTERVENTIONS:
Drug: Ticagrelor 180mg loading dose taken orally, followed by 90mg twice daily (bd) — Ticagrelor 180mg loading dose taken orally, followed by 90mg twice daily (bd)
  Other Names: "Brilinta"

SUMMARY:
A multicenter, single arm, open label, Phase IV study to evaluate safety and to describe the cumulative incidence of major cardiovascular events of Ticagrelor in Taiwanese patients with non ST-segment (a segment in the eletrocardiogram which presents the period when ventricles are depolarized) elevation myocardial infarction

DETAILED DESCRIPTION:
This study will be conducted in approximately 8 investigational centres in Taiwan. It is expected that approximately 100 patients will be enrolled into study treatment. This study is to describe the safety and tolerability of ticagrelor, by assessment of the bleeding events and other serious adverse events (SAEs) during 1year follow up in Taiwanese non ST-elevation myocardial infarction (NSTEMI) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged at least 20 years
3. Patient who is considered as ethnic Taiwanese
4. Index event of non-ST elevation myocardial infarction

Exclusion Criteria:

1. Contraindication or other reason that ticagrelor should not be administered
2. Index event is an acute complication of Percutaneous coronary intervention (PCI)
3. Patient has planned for an urgent coronary artery bypass graft (CABG) within 7 days from the enrolment
4. Oral anticoagulation therapy within 30 days prior to enrolment or cannot be stopped
5. Fibrinolytic therapy in the 24 hours prior to enrolment, or planned fibrinolytic treatment following enrolment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-peng Liu, Ph.D, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (8):
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Niao-Song-Shiang
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Tainan County
  - Research Site, Taipei

REFERENCES:
- See also: RevisedCSP2D5130C00103Redacted_a — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2611&filename=RevisedCSP2D5130C00103Redacted_a.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centres in Taiwan. The first patient was enrolled on 23 April 2015 and the last visit of the last patient took was on 9 February 2017. Informed consent was received for 113 patients
Pre-assignment Details: Out of the patients who provided informed consent 95.6 % (n=108) of the patients received study drug. 8 patients provided informed consent but did not fulfill eligibility criteria, out of whom 5 did not receive treatment and 3 received treatment.
Groups:
- Single Arm: Ticagrelor 90mg twice daily (bd)
Period: Overall Study
Arm/Group | Single Arm
Started | 108
Completed | 99
Not Completed | 9
Not completed — Death | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not hispanic or latino | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fatal/Life-threatening Bleedings
Description: Evaluation of PLATO (PLATelet inhibition and patient Outcomes)-defined fatal/life-threatening bleedings
Time Frame: during 1year follow up with ticagrelor treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Participants
  Fatal/life-threatening bledings | 4

2. Primary Outcome: Number of Participants With Bleeding Events (Major Bleedings)
Description: Evaluation of PLATO (PLATelet inhibition and patient Outcomes)-defined major bleedings
Time Frame: during 1year follow up with ticagrelor treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Participants
  Major bleedings | 7

3. Primary Outcome: Number of Participants With Bleeding Events (Major and Minor Bleedings)
Description: Evaluation of PLATO (PLATelet inhibition and patient Outcomes)-defined major + minor bleedings
Time Frame: during 1year follow up with ticagrelor treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Participants
  Major and minor bleedings | 20

4. Primary Outcome: Number of Participants With Other Serious Adverse Event (SAEs)
Description: Evaluation of serious adverse events other than bleedings
Time Frame: during 1year follow up with ticagrelor treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Participants
  Serious adverse events other than bleeding | 21

5. Primary Outcome: Number of Participants With Major Cardiovascular Events
Description: Evaluation of major cardiovascular events including cardiovascular death, myocardial infarction or stroke
Time Frame: during 1year follow up with ticagrelor treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 108
Participants
  Composite of major cardiovascular events | 6

ADVERSE EVENTS:
Time Frame: On or after the date of first dose and up to and including 7 days following the date of last dose of study medication. 1year if the participant completed treatment according to the study plan. All-cause mortality is collected during 1 year follow-up, including deaths that occur more than 7 days after last dose.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 7/108
Serious Adverse Events (participants affected / at risk) | 23/108
Other Adverse Events (participants affected / at risk) | 45/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=108)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Vascular stent restenosis (General disorders) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=108)
Angina pectoris (Cardiac disorders) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Ecchymosis (Skin and subcutaneous tissue disorders) | 10 (14)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8)
Pyrexia (General disorders) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT02406248/Prot_SAP_000.pdf